CLINICAL TRIAL: NCT04417920
Title: Express Implant Versus Trabeculectomy in a Fibrotic Bleb With Late Failure After Previous Trabeculectomy
Brief Title: Express Implant Versus Trabeculectomy After Late Failure Trabeculectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed Alnagdy, Director, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: late failure trabeculectomy
Record Dates: First submitted 2020-05-21; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Glaucoma
Keywords: Express valve; Failed Trabeculectomy
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy; Mitomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Express implant) (Active Comparator): conjunctival peritomy superior-temporally away from the site of the fibrotic bleb at 12 o'clock, placed on the episclera under the conjunctiva and Tenon's capsule for a contact time of 3 minutes, ,triangular scleral flap , scleral dissection forward to the clear cornea to allow exposure of scleral spur then creation of a pilot hole is fashioned using a sapphire blade (Alcon laboratories,USA) then Express shunt 3 mm long device and external diameter 400 microns was implanted followed by closure of scleral flap and conjunctiva
  Interventions: Procedure: Express implant device
- group II (trabeculectomy) (Active Comparator): Trabeculectomy with Mitomycin-C was done in superior-temporal region away from the fibrotic bleb at 12 o, clock.
  conjunctival peritomy superior-temporally away from the site of the fibrotic bleb at 12 o'clock, placed on the episclera under the conjunctiva and Tenon's capsule for a contact time of 3 minutes, ,triangular scleral flap , scleral dissection forward to the clear cornea to allow exposure of scleral spur then creation of sclerectomy and peripheral iridectomy and closed scleral flab and conjunctiva by nylon 10/0 sutures
  Interventions: Procedure: Express implant device

INTERVENTIONS:
Procedure: Express implant device — Operative technique in group I (Express implant) was as in group II (trabeculectomy) except with no sclerectomy or peripheral iridectomy , the steps included conjunctival peritomy superior-temporally away from the site of the fibrotic bleb at 12 o'clock, placed on the episclera under the conjunctiva and Tenon's capsule for a contact time of 3 minutes, ,triangular scleral flap , scleral dissection forward to the clear cornea to allow exposure of scleral spur then creation of a pilot hole is fashioned using a sapphire blade (Alcon laboratories,USA) then Express shunt 3 mm long device and external diameter 400 microns was implanted followed by closure of scleral flap and conjunctiva.
  While in group II, Trabeculectomy with Mitomycin-C was done in superior-temporal region away from the fibrotic bleb at 12 o, clock.
  Other Names: Trabeculectomy with Mitomycin-C

SUMMARY:
To compare between outcome of Express implant and subscleral trabeculectomy (SST) in management of glaucoma after previous trabeculectomy with a fibrotic bleb.

DETAILED DESCRIPTION:
Trabeculectomy is the main glaucoma surgery. Despite the good decline in intraocular pressure (IOP) that occur rapidly after the procedure, there is still failure occurring due to progressive subconjunctival fibrosis, with associated increased IOP.

If the bleb is revived by needling with adjunctive 5-fluorouracil (5FU) and mitomycin C (MMC) that used intraoperatively for the majority of these cases , the associated rise in IOP was controlled if the revision occured early within the first three months after surgery. But less success occurred if the bleb revision was delayed.

If these interventions fail, alternative approaches include new augmented trabeculectomy or aqueous shunt implantation.

Express shunt allows aqueous to pass from anterior chamber to subconjunctival space like trabeculectomy .Express shunt is a non valved shunt, It has an advantage of less traumatic, less complications, low diffuse bleb and high success rate.

ELIGIBILITY:
Inclusion Criteria:

* elevated intraocular pressure (IOP) with fibrotic bleb despite previous SST since more than 4 months
* follow up 12mo after the second surgery

Exclusion Criteria:

* SST failure other than fibrotic bleb were also excluded
* follow up less than 4mo after the first surgery, and those less than 12mo after the second surgery

Ages: 42 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
change of intra ocular pressure (IOP) | one year follow up
  IOP measured with Goldmann applanation tonometry:
  Complete success in IOP considered as IOP less than 20 mmHg without treatment and a qualified success in IOP considered as IOP less than 20 mmHg with medical treatment and a failure in IOP control considered if IOP more than or equal 20 mmHg after surgery

SECONDARY OUTCOMES:
Visual acuity changes by Decimal | one year follow up
  glaucoma changes follow up
Glaucomatous visual field (VF) changes in median deviation by decibels (dB) | one year follow up
  glaucoma changes follow up
Changes in optic Cup-to-Disc ratio by Volk+90 non-contact lens | one year follow up
  glaucoma changes follow up

CONTACTS AND LOCATIONS:
Overall Officials: Faried Wagdy, Prof., Study Chair — Gamal Abd El Nasr st. - Shebin ElKoum - Menofia
Locations (1):
- Tharwat Mokbel, Al Mansurah, AlDakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740